CLINICAL TRIAL: NCT02624089
Title: Evaluation of the Effect of Intraperitoneal Nebulized Ropivacaine on Morphine Consumption After Laparoscopic Appendectomy in Children. A Prospective, Randomized Double Blind Clinical Trial
Brief Title: Nebulized Analgesia for Laparoscopic Appendectomy Trial
Acronym: NALA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Montreal Children's Hospital of the MUHC (Other)
Responsible Party: Principal Investigator, Robert Baird, Assistant Professor of Pediatric Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-120-PED
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ropivacaine Group (Experimental): This group will receive nebulized ropivacaine 0.5% based on ideal body weight at a dose of 0.5 mg/kg with a maximum total dose of 30 mg. This will be administered once at the onset of pneuomoperitoneum during appendectomy.
  Interventions: Drug: Ropivacaine
- Placebo group (Placebo Comparator): This group will receive placebo (normal saline) based on ideal body weight at a dose of 0.5 mg/kg with a maximum total dose of 30 mg. This will be administered at the onset of pneuomoperitoneum during appendectomy.
  Interventions: Drug: Normal saline
- Non-enrolled group (No Intervention): This group will not receive either intervention (ropivicaine) or placebo (normal saline), but will have primary and secondary endpoints evaluated.

INTERVENTIONS:
Drug: Ropivacaine — Ropivicaine will be administered via in-line nebulization using the Aeroneb Pro™ system
  Other Names: Naropin
  Arms: Ropivacaine Group
Drug: Normal saline — Normal saline will be administered via in-line nebulization using the Aeroneb Pro™ system
  Other Names: 0.9% saline
  Arms: Placebo group

SUMMARY:
The objective of this study is to assess whether the administration of nebulized intra-peritoneal ropivacaine at the onset of surgery, compared with nebulized saline, reduces morphine consumption after laparoscopic appendectomy surgery in children and adolescents.

DETAILED DESCRIPTION:
The laparoscopic approach to pediatric appendectomy is gaining in popularity and has been demonstrated to reduce complications and improve resource utilization. The procedure has a documented association with high postoperative pain intensity, and is associated with substantial pain (pain scores >4 for >60% of the time) in 33% of patients. This is due to surgical manipulation, but also to the intraperitoneal insufflation of carbon dioxide required during laparoscopy which results in in peritoneal stretching, diaphragmatic irritation, changes in intra-abdominal pH as well as retention of insufflation gas in the abdominal cavity after surgery.

Opioid analgesics, especially morphine, are the most common pharmacological option for treating postoperative pain in pediatric patients. Although morphine is generally considered safe to use in pediatric patients, physicians and caregivers often hesitate to prescribe or administer opioids because of the perceived risk of addiction or undesirable side effects. Efforts to mitigate the use of opioids as systemic analgesia after surgery appears warranted. The topical administration of analgesics/anesthetics via the peritoneum is biologically advantageous as intra-abdominal gas insufflation and the resultant increased intra-abdominal pressure generates peritoneal inflammation and neuronal rupture with a linear relationship between abdominal compliance during the procedure and the severity of postoperative pain.

Intraperitoneal nebulization of local a anesthetic agent is a relatively novel approach to pain management after laparoscopy. Intraperitoneal nebulization of local anesthetic allows a uniform dispersion of the agent throughout the peritoneum and combines the analgesic benefits of gas conditioning and local anesthetic instillation. Microvibration-based aerosol humidification devices (i.e. cold nebulization) deliver significant amounts of local anesthetics in the abdominal cavity. Animal studies have confirmed the safety and bioavailability of nebulized ropivicaine in the abdominal cavity. The pharmacokinetics of nebulized ropivacaine 3 mg/kg is similar to that of instilled ropivacaine and maximal ropivacaine concentrations have been found to lie well within safe ranges. Human studies have confirmed favorable pharmacokinetics and pharmacodynamics of nebulized ropivacaine. Peak concentration is attained between 10 and 30 minutes following the end of aerosolized ropivacaine delivery. Aerosolized intraperitoneal local anesthetic is feasible, with ropivacaine concentrations remaining within safe levels.

In previous randomized controlled trials in adults, nebulization of ropivacaine 30 mg with the Aeroneb Pro system either before or after laparoscopic cholecystectomy reduces postoperative pain (effect size - 33% to - 50%) as well as completely prevents shoulder pain compared with nebulization of saline. Patients receiving ropivacaine nebulization consumed significantly less morphine than those in the control group (effects size 40% to -56%). Patients receiving ropivacaine nebulization mobilized quicker than those receiving placebo with a 33% reduction on unassisted walking time after surgery. The duration of analgesia after both pre- and postoperative nebulization (up to 48 hours) was significantly longer than the expected duration of ropivacaine, based on its mechanism of action. No adverse events were reported during the conduct of these trials. Ropivicaine nebulization has also been evaluated in the context of gynecological surgery; patients receiving Ropivacaine 30 mg before or after surgical stimulation reported significantly less postoperative pain (-50%) and consumed significant less morphine (-40%) and walked without assistance than those receiving ropivacaine instillation during the first 24 hours after surgery. Furthermore, the administration of intraperitoneal aerosolized bupivacaine just prior to incising the peri-renal fascia appears to be a simple, effective and low-cost method to reduce postoperative pain in children undergoing laparoscopic pyeloplasty in children.

Given the consistently safe and favorable results documented with adult patients, the working study hypothesis is that the intra-abdominal administration of nebulized ropivacaine immediately before the onset of surgery will reduce post-operative pain and morphine consumption after laparoscopic appendectomy in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 7-18 years old
* ASA Score I (American Society of Anesthesiologists classification) [Appendix 1]: a normal healthy patient.
* ASA Score II (American Society of Anesthesiologists classification): A patient with mild systemic disease
* Patients scheduled for laparoscopic appendectomy surgery
* Uncomplicated appendicitis

  * Hemodynamically stable patient
  * No evidence of appendiceal perforation based on preoperative clinical and imaging assessment
  * Diagnosed to have simple acute appendicitis by intraoperative laparoscopy
* Patients who have provided a written informed assent
* Caregivers who have provided a written informed consent

Exclusion Criteria:

* ASA Score III (American Society of Anesthesiologists classification): A patient with severe systemic disease
* ASA Score IV (American Society of Anesthesiologists classification): A patient with severe systemic disease that is a constant threat to life
* ASA Score V (American Society of Anesthesiologists classification): A moribund patient who is not expected to survive without the operation
* Hemodynamically unstable patient
* Evidence of appendiceal perforation on based on preoperative clinical and imaging assessment
* Perforated or gangrenous appendicitis diagnosed during laparoscopic surgery
* Postoperative admission in an intensive care unit with sedation or ventilatory assistance
* Cognitive impairment or mental retardation
* Progressive degenerative diseases of the CNS
* Seizures or chronic therapy with antiepileptic drugs
* Severe hepatic or renal impairment
* Allergy to one of the specific drugs under study
* Alcohol or drug addiction
* Failure to successfully undergo a laparoscopic appendectomy
* A significant communication problem including language barrier, precluding phone follow up
* Participation in a concomitant research study
* Inability to assure complete follow up
* Failure to acquire informed consent and assent

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Post-operative morphine consumption | During hospital admission (24-48 hours)
  The total dose of Morphine (in mg/kg) and the route of administration received after surgery will be recorded. The oral morphine dose will be converted as 1mg IV= 2mg PO.

SECONDARY OUTCOMES:
Post-operative Pain | During hospital admission (24-48 hours)
  This will be serially evaluated using a Visual Analog Score
Time to unassisted walking | During hospital admission (24-48 hours)
In-hospital length of stay | During hospital admission (24-48 hours)
Postoperative recovery quality | Two weeks after hospital discharge
  This will be evaluated via a standardized telephone questionnaire
Surgeon satisfaction | Immediately after surgery
  this will be evaluated via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert Baird, MDCM MSc, Principal Investigator — Assistant Professor of Pediatric Surgery
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baird R, Ingelmo P, Wei A, Meghani Y, Perez EV, Pelletier H, Auer G, Mujallid R, Emil S, Laberge JM, Puligandla P, Shaw K, Poenaru D. Nebulized analgesia during laparoscopic appendectomy (NALA): A randomized triple-blind placebo controlled trial. J Pediatr Surg. 2019 Jan;54(1):33-38. doi: 10.1016/j.jpedsurg.2018.10.029. Epub 2018 Oct 5. PMID 30366723